CLINICAL TRIAL: NCT02034890
Title: Is Intra - Neobladder Installations of Hyaluronic Acid, Effective in Reducing Neobladder Orthotropic Reconstruction Post-operative Urinary Tract Infections?
Brief Title: Intravesical Instillation of Hyaluronic Acid to Decrease Incidence of Urinary Tract Infection
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty in recruiting patients
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Hanan Goldberg, MD, Rabin Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RMC-7350
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2016-04

CONDITIONS: Urinary Tract Infection
Keywords: orthotopic neobladder; urinary tract infection; intravesical instillation; hyaluronic acid
MeSH Terms: conditions — Urinary Tract Infections | interventions — Hyaluronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hyaluronic acid (Experimental): intravesical instillation of 40 mg of hyaluronic acid at 6 specific time points: 1,2,3 and 4 weeks postoperatively 2 and 3 months postoperatively
  Interventions: Drug: Hyaluronic Acid
- retrospective control patients (No Intervention): retrospective control patients

INTERVENTIONS:
Drug: Hyaluronic Acid — intravesical instillation of 40 mg of hyaluronic acid in 6 specific time points: 1,2,3 and 4 weeks postoperatively (After radical cystectomy and orthotopic neobladder reconstruction) 2 and 3 months postoperatively
  Arms: hyaluronic acid

SUMMARY:
Prospective trial which includes instillation of intravesical hyaluronic acid in an attempt to reduce the incidence of urinary tract infections in patients after orthotopic neobladder reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing radical cystectomy and orthotopic neobladder reconstruction

Exclusion Criteria:

* patients <18 years and unwilling to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
positive urinary culture | 6 months

SECONDARY OUTCOMES:
urinary tract infection | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hanan Goldberg, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Urology department, Rabin Medical Center, Petach Tiqva, Israel